CLINICAL TRIAL: NCT06897540
Title: Screening for Barrett's Esophagus in Patients with Gastroesophageal Reflux Disease: Hospital Based Study
Brief Title: Barrett's Esophagus in Patients with GERD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nervana Nasrat Habib Abd ElMalak, Resident doctor at Assiut University Hospitals, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Barrett's Esophagus
Record Dates: First submitted 2025-03-17; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with GERD (Other): Screening for Barrett's esophagus in patients with GERD by upper endoscopy
  Interventions: Device: Upper endoscopy

INTERVENTIONS:
Device: Upper endoscopy — View mucosa of esophagus with upper endoscope

SUMMARY:
To assess the prevalence and characteristics of BE in patients suffering of chronic GERD symptoms

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is a metaplastic change of the lining of the esophagus with replacement of the normal squamous epithelium with columnar epithelium containing goblet cells. It is the most severe histological consequence of chronic gastroesophageal reflux and predisposes to the development of adenocarcinoma of the esophagus (Spechler SJ et al., 2001).

BE develops when metaplastic columnar mucosa replaces the normal esophageal squamous epithelium of the esophagus in response to damage caused by gastroesophageal reflux . The columnar-lined esophagus contains a mosaic of 3 different cell types: gastric fundic type epithelium, junctional cardiac epithelium, and specialized columnar epithelium with intestinal type goblet cells. Most professional guidelines from around the world agree that a diagnosis of BE requires the presence of Intestinal Metaplasia (IM) because of an increased risk of Esophageal Adenocarcinoma (EAC )associated with IM, although guidelines from the British Society of Gastroenterology and the Asia Pacific region do not require this (Shaheen NJ et al., 2022).

The poor prognosis of EAC has focused interest on BE. Identification of BE with treatment of dysplasia is important to prevent invasive cancer. On the other hand, gastroesophageal reflux disease (GERD) has been associated with an increased risk of BE. Despite recommendations against population-based screening, the majority of guidelines recommend considering screening of chronic GERD patients. However, 50% of EAC patients report no previous GERD (Marques de Sá I et al., 2020).

Current guidelines for the diagnosis and treatment of GERD state that empiric therapy should be given to patients with typical heartburn, and it is recommended that patients with chronic GERD symptoms undergo upper endoscopy (Sampliner R et al., 2005).

.The columnar metaplasia in BE causes no symptoms. Thus, patients are seen initially for symptoms of the associated GERD, such as heartburn and regurgitation. Endoscopically obvious BE can be seen in approximately 10% of patients who have endoscopic examinations for symptoms of GERD. However, approximately 25% of patients have no esophageal symptoms (Winters C Jr et al., 1987).

BE is usually discovered during endoscopic examination of middle-aged and older adults whose mean age at the time of diagnosis is approximately 55 years (Spechler SJ et al., 1996).

BE is best described by using the validated Prague criteria that includes both the circumferential and maximal extent of the columnar epithelium in the esophagus and the location of the proximal margin of the gastric folds and the diaphragmatic hiatus (Shaheen NJ et al., 2022). BE is associated with several risk factors. These include chronic reflux symptoms (defined as weekly symptoms for 5 or more years), male sex, age greater than 50 years, smoking, white race, central obesity, and family history. The prevalence in those with GERD and 1 additional risk factor was, however, substantially higher than GERD alone (12.2%). In addition, a positive linear relationship was also shown between the number of risk factors and BE prevalence, with each additional risk factor increasing the prevalence of BE by 1.2% (Shaheen NJ et al., 2022).

ELIGIBILITY:
Inclusion Criteria:

Adults diagnosed with GERD based on clinical symptoms and/or 24-hour pH monitoring or esophageal manometry.

Patients willing to undergo endoscopic examination

Exclusion criteria: Patients with a history of esophageal cancer.

Patients with other esophageal diseases, such as eosinophilic esophagitis, infections, or motility disorders.

Patients who are unable to consent or participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
To assess the prevalence and characteristics of BE in patients suffering of chronic GERD symptoms. | Assessment of patients with GERD take about 2 weeks
  To assess the prevalence and characteristics of BE in patients suffering of chronic GERD symptoms.
  To evaluate demographic and clinical risk factors associated with BE in GERD patients.
  To assess the clinical features of GERD in patients who develop BE. To investigate the diagnostic methods used to detect BE in clinical settings. To assess the relationship between chronicity of GERD and development of BE.

IPD SHARING:
Plan to Share IPD: No
Only patients who will be discovered having Barrett's esophagus will their IPD ba shared